CLINICAL TRIAL: NCT02902627
Title: Pain in Oncolgy: Evaluation of a Non Invasive Monitoring Device (ANI). A Monocentric Prospective Study
Acronym: ANIONCO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2011/64; 2011-A01559-32 (Other: ANSM)
Record Dates: First submitted 2016-09-13; First posted 2016-09-16 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Pain; Cancer
MeSH Terms: conditions — Pain; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Metastatic cancer (Experimental)
  Interventions: Device: Non Invasive Monitoring Device (ANI)

INTERVENTIONS:
Device: Non Invasive Monitoring Device (ANI) — Pain measure by ANI monitor and with visual analogical scale

SUMMARY:
l'ANI (Analgesia Nociception Index

The main objective of the research is to estimate the Analgesia Nociception Index (ANI) as a parameter giving the possibility of measuring the pain in painful metastatic cancer. The parameter ANI is compared with visual analogical scale (VAS) score.

ELIGIBILITY:
Inclusion Criteria:

* more than 18 years, -no legal protection, -
* life expectancy is considered over 3-months
* not receiving of béta-blocking,
* Having a rhythm sinusal without extrasystole
* benefiting from a coverage by a social security system

Exclusion Criteria:

* Pace-Maker
* Diabetes mellitus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-08; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Comparison of the ANI parameter with the VAS | 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Marc Fischler, Principal Investigator — Hopital Foch
Locations (1):
- Hopital Foch, Suresnes, France

IPD SHARING:
Plan to Share IPD: No